CLINICAL TRIAL: NCT03550053
Title: A 3D Analysis of Mandibular Plating Strategies in Oromandibular Reconstruction: A Single- Blinded Randomized Controlled Trial.
Brief Title: A 3D Analysis of Mandibular Plating Strategies in Oromandibular Reconstruction.
Acronym: 3Dplating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 16-5984
Record Dates: First submitted 2017-11-14; First posted 2018-06-08 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with head and neck cancer, specifically requiring surgery to their mandible.
Who Masked: Participant
Masking Description: Patient will not know which group they are randomized to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intraoperative plate bending (Active Comparator): Plate will be bent intraoperatively, which is the standard of care, for this surgery
  Interventions: Device: 3D mandibular plate
- Preoperative plate bending (Active Comparator): A 3D printed model of the patient's mandible will be used to bend the plate preoperatively by the surgeon. The pre-bent plate will be brought into the operating room on the day of surgery.
  Interventions: Device: 3D mandibular plate

INTERVENTIONS:
Device: 3D mandibular plate — Patients will be randomly assigned to either have the mandibular plate bent before their surgery, using a 3D model of their mandible or have the mandibular plate bent during their surgery, which is standard of care.

SUMMARY:
Reconstruction of the mandible commonly employs the use of metal plates to provide a framework for placement of bone grafts. The standard approach to reconstruction involves bending these plates to the mandible intraoperatively. A novel technique involves bending plates to three dimensional (3D) printed models of the mandible prior to surgery. No study has performed a quantitative analysis and comparison of these two different strategies. The purpose of this study is to compare reconstructive plating strategies (preoperative versus intraoperative bending) for mandibular reconstruction using 3D quantitative analysis. Preoperative diagnostic CT scans of the head/neck of 20 patients scheduled to undergo mandibular reconstruction will be obtained and imported into 3D modeling software. A computer based 3D reconstructed mandible will be printed. Simulated reconstruction will be replicated by contouring mandibular reconstruction plates to each model. The plates will be marked, sterilized and brought to the operating room on the day of surgery. Each patient will be randomized to either preoperative (n=10) or intraoperative (n=10) plate bending groups. The group will be revealed to the primary surgeon on the day of surgery and the patient will either be fit with the plate bent preoperatively or will undergo fitting with a plate bent intraoperatively. Following reconstruction of the mandible, the patient will undergo intraoperative cone beam scanning. Using scans performed pre- and post-mandibular reconstruction, the 3D simulated mandibles will be compared based on the position of the mandibular condyle within the Temporomandibular Joint. In addition, the percentage of surface area contact between the plate and mandible and the postoperative occlusion attained will be determined and compared between groups. It is expected that the preformed plates will have improved contact surface area, and better achieve pre-reconstruction occlusion when compared to plates bent intraoperatively.

DETAILED DESCRIPTION:
Patients will be identified through attendance at the Wharton Head and Neck Clinic at Princess Margaret Hospital or attendance at the Toronto General Hospital Otolaryngology - Head & Neck Surgery clinic as requiring resection of mandibular pathology and subsequent reconstruction with bony free flap. Chart review (electronic) of these patients will be performed to obtain demographic information and factors such as tumor type, site, stage and prior treatment. Data will be obtained from CT scans to create 3D models, including anatomic parameters required for 3D printing of the mandible. Following reconstruction, a number of variables will be collected (i.e. position of the mandibular condyle within the temporomandibular joint, percentage of surface area contact between the plate and bone, type of occlusion/bite and degree of conformance). All of this data will be stored in a password protected Excel spreadsheet located on a secure University Health Network computer. Twenty participants will be enrolled into this study and randomized to one of two groups: intraoperative plate bending (n=10) or preoperative plate bending (n=10) using a 3D printed model. While the participant can be blinded to the strategy that will be pursued, the surgeon performing the reconstruction will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing planned resection with osseous free flap reconstruction of the mandible
* Pathology limited to unilateral involvement of the mandible from the angle to the mandibular symphysis (lateral defects)

Exclusion Criteria:

* Patients under age 18
* Prior reconstruction of the mandible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Jaw contour | 1 week after surgery
  Contour of the mandible will be measured using the pre and post-op CT images. A comparison will be made between the sets of images to determine which strategy of reconstruction (pre-bent plate or intraoperative bent plate) better recreates the native contours of the mandible.

SECONDARY OUTCOMES:
Change in Jaw occlusion | 1 week after surgery
  Occlusion of the mandible will be measure using the pre and post-op CT images. A comparison will be made between the sets of images to determine which strategy of reconstruction (pre-bent plate or intraoperative bent plate) better recreates the natural bite/occlusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada